CLINICAL TRIAL: NCT04613245
Title: Health-Related Quality of Life of Patients With Asthma and Its Associated Factors During the Pandemic of COVID-19
Brief Title: Health-Related Quality of Life of Patients With Asthma During the Pandemic of COVID-19
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Naglaa Fathy Afifi Youssef, Assistant professor, Cairo University
Other Study IDs: Serial 39-2020
Record Dates: First submitted 2020-10-29; First posted 2020-11-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Asthma Chronic; Bronchial Asthma
Keywords: Quality of life; Health related quality of life; patient reported outcome; Asthma; COVID-19
MeSH Terms: conditions — Asthma; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with asthma

SUMMARY:
Nowadays, the COVID-19 epidemic causes stress not only to healthy people but also to people with unhealthy conditions. Excess psychological stress (either in quality, quantity, frequency, and/or duration) could push susceptible individuals to ultimately develop clinical asthma. Depression was significantly associated with asthma interference with daily activities, breathlessness, night symptoms, use of bronchodilators, and poor compliance with medical treatment.

Covid-19 pandemic induced the countries around the world to require from its citizens not to ask for health care support rather than in emergency situations and through utilizing telemedicine. This action aims to control spreading the infection with viruses as well as to reduce the workload on the healthcare providers.

Although asthma is not listed as one of the chronic conditions that might complicate coronavirus infections, asthma people might have a high-stress level that might induce their asthma attack which consequentially reflects on their quality of life. People with asthma have a unique experience rather than people with other health conditions during COVID-19.

Patients with asthma experience a lot of stressors that might induce asthma and impaired their HRQOL such as overuse of antiseptic substances, stay home with a sedentary lifestyle, the sudden shift to telemedicine, and electronic work from home. Also, as a result of the similarity of asthma symptoms with coronavirus symptoms, the patient might have a continuous sense of uncertainty that s/he is infected with the COVID-19 virus, and this suspicion can increase the psychological overburden on these patients.

Therefore, all these stressors should be evaluated to recognize their health needs and the kind of social and health support that should be provided to them during the pandemic time. Also, Identifying the predictors of HRQOL among patients with asthma during the pandemic of COVID-19 is urgently required.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disease of the lower respiratory tract which derives from a combination of genetic predisposition with environmental exposure to several factors. It is a chronic respiratory disease that results in morbidity, mortality, and impaired health-related quality of life (HRQoL). It is estimated that 334 million people have asthma worldwide.

Nowadays, the COVID-19 epidemic causes stress not only to healthy people but also to people with unhealthy conditions. Excess psychological stress (either in quality, quantity, frequency, and/or duration) could push susceptible individuals to ultimately develop clinical asthma. Depression was significantly associated with asthma interference with daily activities, breathlessness, night symptoms, use of bronchodilators, and poor compliance with medical treatment.

Covid-19 pandemic induced the countries around the world to require from its citizens not to ask for health care support rather than in emergency situations and through utilizing telemedicine. This action aims to control spreading the infection with viruses as well as to reduce the workload on the healthcare providers.

Although asthma is not listed as one of the chronic conditions that might complicate coronavirus infections, asthma people might have a high-stress level that might induce their asthma attack which consequentially reflects on their quality of life. People with asthma have a unique experience rather than people with other health conditions during COVID-19.

Patients with asthma experience a lot of stressors that might induce asthma and impaired their HRQOL such as overuse of antiseptic substances, stay home with a sedentary lifestyle, the sudden shift to telemedicine, and electronic work from home. Also, as a result of the similarity of asthma symptoms with coronavirus symptoms, the patient might have a continuous sense of uncertainty that s/he is infected with the COVID-19 virus, and this suspicion can increase the psychological overburden on these patients.

Therefore, all these stressors should be evaluated to recognize their health needs and the kind of social and health support that should be provided to them during the pandemic time. Also, Identifying the predictors of HRQOL among patients with asthma during the pandemic of COVID-19 is urgently required.

A cross-sectional analytical design will be utilized.

The study participants will be adults (18 years or older) who have been diagnosed with bronchial asthma or pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Participant's age: 18 years or older
* medically diagnosed with bronchial asthma

Exclusion Criteria:

* not medically diagnosed with asthma by a physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study participants will be adults who have been diagnosed with bronchial asthma or pulmonary disease.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire (ACQ) | One week
  ACQ has a multidimensional construct assessing symptoms (5 items--self-administered) and rescue in bronchodilator use (1 item-self-administered), and FEV1% (1 item) completed by clinic staff, but it will not be applied in the current study as it will be difficult to be self-reported by the participants. 7-point scale (0=no impairment, 6= maximum impairment for symptoms. Scores range between 0 (totally controlled) and 6 (severely uncontrolled).

SECONDARY OUTCOMES:
Mini Asthma Quality of Life Questionnaire | two weeks
  The MiniAQLQ will be utilized to investigate the HRQoL of the participants. The Mini AQLQ-S has 15 questions that gives an overall summary index and four domains: activity limitation, symptoms, emotional function, and environmental stimuli. The questions all refer to the "last two weeks" and use seven Likert-type response options e.g., seven response options ranging from "all of the time" to "none of the time".

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa FA Youssef, PhD, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided